CLINICAL TRIAL: NCT02897973
Title: Spinal Loads During Activities of Daily Living: Influences of Unilateral Lower-limb Amputation
Brief Title: The Impact of Unilateral Lower Limb Amputation on Spinal Loads
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Babak Bazrgari, PhD, Principal Investigator, University of Kentucky
Other Study IDs: R03HD086512-01A1 (NIH)
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
Keywords: Spinal loads; Trunk muscle force; Computational modeling; Unilateral lower limb amputation
MeSH Terms: conditions — Low Back Pain | interventions — Activities of Daily Living

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Transtibial lower limb amputation: unilateral amputation below knee resulting from traumatic injuries (with no upper-extremity amputations), evaluation took place at least 6 months post-injury, no assistive device use (e.g., canes, walkers, crutches), no other documented injuries, such as musculoskeletal impairments in the contralateral limb, neurologic disorder or traumatic brain injury that would affect gait and movement.
  Interventions: Other: Activity of daily living
- Transfemoral lower limb amputation: unilateral amputation above knee resulting from traumatic injuries (with no upper-extremity amputations), evaluation took place at least 6 months post-injury, no assistive device use (e.g., canes, walkers, crutches), no other documented injuries, such as musculoskeletal impairments in the contralateral limb, neurologic disorder or traumatic brain injury that would affect gait and movement.
  Interventions: Other: Activity of daily living
- Controls: Able-bodied individuals without amputation
  Interventions: Other: Activity of daily living

INTERVENTIONS:
Other: Activity of daily living — walking, sitting-to-standing and standing-to-sitting, stairs ascending and descending

SUMMARY:
The prevalence of low back pain among persons with unilateral lower limb amputation is significantly higher than the rate experienced by the general public. Chronic pain, including low back pain, limits functional independence and negatively impacts quality of life. As such, this project will investigate the role of a biomechanical casual pathway in the development of low back pain; to do this, the investigators will explore the relationship between the adopted neuromuscular patterns post-amputation to perform activities of daily living and the risk of developing spinal tissue damage.

DETAILED DESCRIPTION:
Despite the higher prevalence of low back pain (LBP) among persons with unilateral lower limb amputation (ULLA) compared to able-bodied individuals, relatively little is known about the fundamental mechanisms underlying this condition. This research represents a first step toward investigating lower back biomechanics using advanced computational modeling techniques to inform the future design of effective interventions for LBP. Specifically, the impact of trunk neuromuscular patterns adopted by persons with ULLA while performing activities of daily living on spinal loads and the risk of spinal tissue damage will be investigated. This will be achieved via secondary biomechanical analyses of a large set of high-quality kinematics data obtained from individuals with and without ULLA performing the following tasks: 1) walking at self-selected and controlled speeds, 2) sit-to-stand and stand-to-sit, and 3) stairs-up and stairs-down. The central hypothesis is that, compared to able-bodied individuals, trunk movement strategies adopted by persons with ULLA to cope with physical demands of common daily activities are associated with a complex pattern of internal muscle forces that result in larger loads on the spine and a higher probability for spinal tissue damage. Investigators' dataset draws from the Biomechanics Laboratory at Walter Reed National Military Medical Center (WRNMMC) which has unprecedented access to a large population of service members with ULLA. Using this unique database, investigators will implement their novel finite element modeling approach to estimate the internal muscle forces (i.e., adopted neuromuscular patterns) needed to perform daily physical activities on the basis of satisfying equilibrium and stability across the entire lumbar spine. Completion of this project will enable the investigators to determine differences in muscle recruitment, as well as the resultant effects on spinal loads and the risk of spinal tissue damage, between persons with and without ULLA. Hence, this pilot project is expected to establish the initial groundwork for future research involving the design of highly specific interventions aimed at trunk neuromuscular behaviors during post-amputation rehabilitation to lessen adverse effects on lower back biomechanics and the potential for LBP.

ELIGIBILITY:
Inclusion Criteria:

For individuals with amputation

* unilateral amputation resulting from traumatic injuries (with no upper-extremity amputations)
* evaluation took place at least 6 months post-injury
* no assistive device use (e.g., canes, walkers, crutches)

For controls:

* able-bodied individuals without amputation
* to be matched with group with ampuation on the basis of anthropometric measure

Exclusion Criteria:

For individuals with amputation:

* musculoskeletal impairments in the contralateral limb
* neurologic disorder or traumatic brain injury that would affect gait and movement
* pain levels greater than 3 out of 10 on a visual analog scale
* a history of spinal pathologies/LBP prior to injury.

For controls

* a history of spinal pathologies/LBP

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project involves secondary analyses of existing data and so will not include a subject recruitment process. Kinematics data collected at Walter Reed National Military Medical Center will be used for estimation of internal muscle forces and the resultant spinal loads and the probability of spinal tissue damage during several basic activities of daily living using a computational model of the lower back. Following an initial assessment, the investigators estimate the following available sample sizes for each activity of daily living: (transfemoral-TFA, transtibial-TTA, and Controls-CTL ) 1) level ground walking at four different speeds (nTFA= 57, nTTA= 53, nCTL= 32), 2) sitting-to-standing and standing-to-sitting (nTFA= 29, nTTA= 20, nCTL= 15), and 3) stair ascending and descending tasks (nTFA= 18, nTTA= 20, nCTL= 15).
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maximum value of summation of predicted forces in all trunk muscles | At least 6 months post-injury
  All outcome measures are obtained from computational simulation of data collected in previous studies.
Maximum spinal load at the lowest level of lumbar spine | At least 6 months post-injury
  All outcome measures are obtained from computational simulation of data collected in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Bazrgari, PhD, Principal Investigator — University of Kentucky